CLINICAL TRIAL: NCT03154619
Title: Efficacy of TR 987, Beta-1,3-1,6-D-glucan, in the Treatment of Chronic Venous Insufficiency Ulcers: a Two-arm, Double-blind, Placebo-controlled, Randomized Controlled Trial.
Brief Title: Efficacy of TR 987, Beta-1,3-1,6-D-glucan, in the Treatment of Chronic Venous Insufficiency Ulcers
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SerenaGroup, Inc. (Network)
Collaborators: TR Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BG001
Record Dates: First submitted 2017-05-12; First posted 2017-05-16 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer | interventions — beta-Glucans

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TR987 (Active Comparator): This group will receive twice-weekly applications of 0.1% TR 987 in a gel base plus SoC for the first 4 weeks, then once weekly applications for the remaining 8 weeks of the trial.
  Interventions: Drug: 0.1% TR 987
- Placebo (Placebo Comparator): This group will receive twice-weekly applications of placebo gel base plus SoC for the first 4 weeks, then once weekly applications for the remaining 8 weeks of the trial.
  Interventions: Drug: Placebo gel

INTERVENTIONS:
Drug: 0.1% TR 987 — TR 987 0.1%
  Other Names: Beta glucan
  Arms: TR987
Drug: Placebo gel — Placebo gel twice weekly for 4 weeks, then once weekly for 8 weeks. Gel will be applied to cover the wound cavity and wound surface to a thickness of 5 mm.
  Arms: Placebo

SUMMARY:
The safety and efficacy of beta glucan products, and specifically TR 987, in the treatment of chronic venous insufficiency ulcers has been established. This study is designed to determine the most efficient method of treatment.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled study to evaluate the effectiveness of TR 987 gel. It is a two-arm, design: One group will receive twice-weekly applications of 0.1% TR 987 in a gel base plus SoC for the first 4 weeks. The other group will receive twice-weekly applications of placebo gel base plus SoC for the same period of time. After 4 weeks, both groups will receive once weekly applications of their assigned treatment for the remaining 8 weeks of the trial. The Standard of Care therapy in this study is multi-layer compression therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years old
2. Female subjects are not pregnant or breastfeeding.
3. Study ulcer has been present for at least one month and has undergone more than 2 weeks, but less than 12 months of continuous high-strength compression with less than 40% healing.
4. Study ulcer is a minimum of 2.0 cm2 and a maximum of 20.0 cm2, extending through the full thickness of the skin, but not down to muscle, tendon, or bone at the randomization visit.
5. Study ulcer has a clean, granulating base with minimal adherent slough at the randomization visit.
6. If more than one ulcer is present on the same leg, they must be more than 2 cm apart and only the larger ulcer will be included in the study.
7. Adequate arterial flow, as measured by an Ankle Brachial Pressure Index (ABI) of greater than 0.75. (Calculations will be made using measurements from both posterior tibial and dorsalis pedis arteries, as well as both arms) and/or Skin Perfusion Pressure (SPP) >30.
8. Subject understands and is willing to participate in the clinical study and can comply with weekly visits and the follow-up regimen.
9. Patient understands and is willing to participate in the clinical study and can comply with weekly visits and the follow-up regimen.
10. Patient has read and signed the IRB/IEC approved Informed Consent Form before screening procedures are undertaken.

Exclusion Criteria:

1. Study ulcer deemed by the Investigator to be caused by a medical condition other than venous insufficiency.
2. Study ulcer exhibits clinical signs and symptoms of infection.
3. Study ulcer requires enzymatic debridement during the study.
4. Study ulcer has undergone 12 or more months of continuous high-strength compression therapy over its duration.
5. Study ulcer is less than 2.0 cm2 or greater than 20.0 cm2.
6. Study ulcer extends more than 50% below the malleolus.
7. Study ulcer is treated with a topical antibiotic during the screening phase.
8. Study ulcer has been treated with tissue engineered material (e.g., Apligraf® or Dermagraft®) or other scaffold materials (e.g., Oasis or Matristem) within 30 days prior to the TV1 Randomization visit.
9. Study ulcer requiring negative pressure wound therapy or hyperbaric oxygen during the course of the trial.
10. History of radiation at the study ulcer site.
11. Study ulcer decreases in area by 30% or more during the 14 days screening period.
12. Subjects who are unable to understand the aims and objectives of the trial or has a known history of poor adherence with medical treatment.
13. Presence of any condition(s) that seriously compromises the subject's ability to complete this study.
14. All females of childbearing potential who are not using a highly effective method of birth control (failure rate less than 1% per year), such implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence or vasectomized partner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-04-04 (Actual); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Time to complete wound closure | 12 weeks

SECONDARY OUTCOMES:
Percentage of subjects with complete ulcer healing | 12 weeks
Change in ulcer size | 4 weeks
Change in ulcer size | 12 weeks
Incidence of adverse events | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Serena, MD, Principal Investigator — SerenaGroup, Inc.
Locations (9):
- United States (9):
  - New Hope Podiatry Clinic, Los Angeles, California
  - Barry University Clinical Research, North Miami Beach, Florida
  - Royal Research Corp, Pembroke Pines, Florida
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Cleveland Foot and Ankle Clinic, Cleveland, Ohio
  - The Foot and Ankle Wellness Center, Ford City, Pennsylvania
  - Armstrong County Memorial Hospital, Kittanning, Pennsylvania
  - SerenaGroup Research Institute, Pittsburgh, Pennsylvania
  - Martin Foot and Ankle, York, Pennsylvania

IPD SHARING:
Plan to Share IPD: No